CLINICAL TRIAL: NCT00670449
Title: An Extension of the 6-month, Double-blind, Randomized, Placebo-controlled, Parallel-group, Multicenter Study Comparing Efficacy and Safety of FTY720 0.5 mg and 1.25 mg Administered Orally Once Daily in Patients With Relapsing Multiple Sclerosis
Brief Title: An Extension Study of the Efficacy and Safety of Fingolimod (FTY720) in Patients With Relapsing Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CFTY720D1201E1
Record Dates: First submitted 2008-04-28; First posted 2008-05-01 (Estimated); Results first posted 2013-09-04 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-06

CONDITIONS: Multiple Sclerosis
Keywords: FTY720; multiple sclerosis; MS
MeSH Terms: conditions — Multiple Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Fingolimod 0.5 mg (Experimental): Patients who received fingolimod 0.5 orally once daily in the core study continued on the same dose in this extension study.
  Interventions: Drug: Fingolimod
- Fingolimod 1.25 mg (Experimental): Patients who received fingolimod 1.25 mg orally once daily in the core study continued on the same dose in this extension study.
  Interventions: Drug: Fingolimod
- Placebo-fingolimod (Experimental): Patients who were randomized to placebo in the core study were re-randomized to either fingolimod 0.5 or 1.25 mg (1:1) orally once daily in this extension study.
  Interventions: Drug: Fingolimod

INTERVENTIONS:
Drug: Fingolimod — Fingolimod was supplied in capsules.
  Other Names: Gilenya; Imsera

SUMMARY:
This study was an extension study of NCT00537082. This study was designed to evaluate the efficacy and safety of long-term administration of 0.5 mg or 1.25 mg of fingolimod (FTY720) to relapsing multiple sclerosis.

DETAILED DESCRIPTION:
A decision was made to switch all patients on fingolimod 1.25 mg/day to fingolimod 0.5 mg/day in an amendment to the study protocol. The study became open-label with all patients receiving fingolimod 0.5 mg/day on 22 Feb 2010.

The efficacy data for Months 0-6 in this study report is from the core study NCT00537082.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed 6 months of treatment with the study drug and the Month 6 visit in the core study NCT00537082.
* Females of childbearing potential who have a negative pregnancy test in the core study NCT00537082.

Exclusion Criteria:

* Patients who permanently discontinued study drug treatment prior to the Month 6 visit in the core study NCT00537082.

Other protocol-defined inclusion/exclusion criteria applied to the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 143 (Actual)
Dates: Start 2008-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Japan, Principal Investigator — 81-3-3797-8748
Locations (15):
- Japan (15):
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Ehime
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Gunma
  - Novartis Investigative Site, Hyōgo
  - Novartis Investigative Site, Ibaraki
  - Novartis Investigative Site, Kanagawa
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Morioka
  - Novartis Investigative Site, Niigata
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Sapporo
  - Novartis Investigative Site, Tochigi
  - Novartis Investigative Site, Tokyo
  - Novartis Investigative Site, Wakayama

REFERENCES:
- [Derived] Saida T, Itoyama Y, Kikuchi S, Hao Q, Kurosawa T, Ueda K, Auberson LZ, Tsumiyama I, Nagato K, Kira JI. Long-term efficacy and safety of fingolimod in Japanese patients with relapsing multiple sclerosis: 3-year results of the phase 2 extension study. BMC Neurol. 2017 Jan 28;17(1):17. doi: 10.1186/s12883-017-0794-5. PMID 28129749
- [Derived] Kira J, Itoyama Y, Kikuchi S, Hao Q, Kurosawa T, Nagato K, Tsumiyama I, von Rosenstiel P, Zhang-Auberson L, Saida T. Fingolimod (FTY720) therapy in Japanese patients with relapsing multiple sclerosis over 12 months: results of a phase 2 observational extension. BMC Neurol. 2014 Jan 29;14:21. doi: 10.1186/1471-2377-14-21. PMID 24475777

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo-fingolimod 0.5 mg; Placebo-fingolimod 1.25 mg: Patients who were randomized to placebo in the core study were re-randomized to either fingolimod 0.5 or 1.25 mg (1:1) orally once daily in this extension study.
Period: Overall Study
Arm/Group | Fingolimod 0.5 mg | Fingolimod 1.25 mg | Placebo-fingolimod 0.5 mg | Placebo-fingolimod 1.25 mg
Started | 47 | 46 | 27 | 23
Switched to 0.5mg (Open Label) | 45 | 41 (Following protocol amendment, study became open-label with all patients receiving FTY720 0.5 mg/day) | 23 | 17 (Following protocol amendment, study became open-label with all patients receiving FTY720 0.5 mg/day)
Completed | 38 | 36 | 18 | 15
Not Completed | 9 | 10 | 9 | 8
Not completed — Adverse Event | 6 | 2 | 8 | 5
Not completed — Protocol Deviation | 1 | 2 | 0 | 1
Not completed — Administrative Problems | 0 | 2 | 0 | 1
Not completed — Subject Withdrew Consent | 0 | 2 | 0 | 1
Not completed — Unsatisfactory Therapeutic Effect | 2 | 0 | 1 | 0
Not completed — Abnormal Laboratory Value(s) | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fingolimod 0.5 mg | Fingolimod 1.25 mg | Placebo-fingolimod 0.5 mg | Placebo-fingolimod 1.25 mg | Total
Number analyzed (Participants) | 47 | 46 | 27 | 23 | 143
Age Continuous [Mean (Standard Deviation); unit: years] | 34.9 (8.95) | 35.7 (8.81) | 34.2 (9.08) | 35.5 (8.44) | 35.1 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 31 | 19 | 14 | 97
  Male | 14 | 15 | 8 | 9 | 46

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Free of Gd-enhanced T1 Weighted Magnetic Resonance Imaging (MRI) Lesions
Description: To ensure consistency, MRI scans were evaluated centrally at the Institute of Neurotherapeutics in Kyoto, Japan. After checking the scans for completeness and quality, all scans were analyzed by blinded readers (experienced neurologists). The number of Gd-enhanced T1 weighted MRI lesions were counted and recorded. Lesions expanding through several slices were counted as only 1 lesion.
Time Frame: Months 6, 9, 12, 18, 24, 36, and 48
Population: Core full analysis set (FAS): All patients who were randomized in the core study and received at least 1 dose of core study drug. The study became open-label with all patients receiving FTY720 0.5 mg/day (by 22-Feb- 2010). (approximately 22 months before study completion)
Measure: Number; unit: Percentage of patients
Groups:
- Placebo-fingolimod: Patients randomized to placebo in the Core study. These patients were either subsequently re-randomized to FTY720 (either 1.25 mg or 0.5 mg) in the Extension study, or did not enter the Extension study.
Arm/Group | Fingolimod 0.5 mg | Fingolimod 1.25 mg | Placebo-fingolimod
Number analyzed (Participants) | 57 | 54 | 57
Percentage of patients
  Month 6 (N=44, 48, 50) | 88.6 | 97.9 | 58.0
  Month 9 (N=44, 39, 41) | 90.9 | 94.9 | 92.7
  Month 12 (N=44, 42, 36) | 97.7 | 97.6 | 88.9
  Month 18 (N=42, 40, 37) | 92.9 | 92.5 | 94.6
  Month 24 (N=38, 39, 33) | 94.7 | 94.9 | 90.9
  Month 36 (N=25, 21, 22) | 92.0 | 85.7 | 90.9
  Month 48 (N=3, 4, 1) | 100.0 | 75.0 | 100.0

2. Secondary Outcome: Percentage of Patients Free of New or Newly Enlarged T2 Weighted MRI Lesions
Description: To ensure consistency, MRI scans were evaluated centrally at the Institute of Neurotherapeutics in Kyoto, Japan. After checking the scans for completeness and quality, all scans were analyzed by blinded readers (experienced neurologists). The number of new or newly enlarged T2 weighted MRI lesions were counted and recorded. New lesions were identified by comparing each lesion with previous scans. Lesions expanding through several slices were counted as only 1 lesion.
Time Frame: Months 0-3, 3-6, 6-9, 9-12, 12-18, 18-24, 24-36,36-48, and 48 to the end of the study (up to 4 years)
Population: Core full analysis set(FAS): All patients who were randomized in the core study and received at least 1 dose of core study drug. Study became open-label with all patients receiving FTY720 0.5 mg/day. The study became open-label with all patients receiving FTY720 0.5 mg/day (by 22-Feb-2010). (approximately 22 months before study completion)
Measure: Number; unit: Percentage of patients
Arm/Group | Fingolimod 0.5 mg | Fingolimod 1.25 mg | Placebo-fingolimod
Number analyzed (Participants) | 57 | 54 | 57
Percentage of patients
  Month 0 to 3 (N=49, 50, 51) | 69.4 | 60.0 | 45.1
  Month 3 to 6 (N=43, 47, 48) | 86.0 | 91.5 | 43.8
  Month 6 to 9 (N=44, 39, 40) | 88.6 | 92.3 | 70.0
  Month 9 to 12 (N=44, 42, 35) | 93.2 | 95.2 | 85.7
  Month 12 to 18 (N=43, 40, 37) | 88.4 | 90.0 | 91.9
  Month 18 to 24 (N=39, 39, 33) | 94.9 | 92.3 | 87.9
  Month 24 to 36 (N=25, 21, 22) | 92.0 | 90.5 | 90.9
  Month 36 to 48 (N=3, 4, 1) | 100.0 | 100.0 | 100.0
  Month 48 to end of study (N=3, 3, 1) | 100.0 | 100.0 | 100.0

3. Secondary Outcome: Aggregate Annualized Relapse Rate (ARR) Based on Confirmed Relapses
Description: The ARR was defined as the total number of relapses for all patients in the treatment arm / total number of days in the study for all patients in the treatment arm for the specific period of time × 365.25. General definition of relapse: Appearance of a new neurological abnormality or worsening of previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from the onset of a preceding clinical demyelinating event. The abnormality must be present for at least 24 hours and occur in the absence of fever (< 37.5°C) or infection. A relapse was to be confirmed by a neurologist trained on the Expanded Disability Status Scale (EDSS). A relapse must be accompanied by an increase of at least half a step (0.5) on the EDSS or an increase of 1 point on 2 different Functional Systems (FS) of the EDSS or 2 points on 1 of the FS (excluding Bowel/Bladder or Cerebral FS).
Time Frame: Months 0-6, 6-12, 12-24, 24-36, 36-48, and 48 to the end of the study (up to 4 years)
Population: as for outcome 1
Measure: Number; unit: Relapses per year
Arm/Group | Fingolimod 0.5 mg | Fingolimod 1.25 mg | Placebo-fingolimod
Number analyzed (Participants) | 57 | 54 | 57
Relapses per year
  Month 0 to 6 (N=57, 54, 57) | 0.539 | 0.404 | 1.131
  Month 6 to 12 (N=47, 46, 50) | 0.227 | 0.284 | 0.232
  Month 12 to 24 (N=44, 43, 39) | 0.166 | 0.223 | 0.222
  Month 24 to 36 (N=41, 40, 34) | 0.191 | 0.058 | 0.162
  Month 36 to 48 (N=28, 23, 23) | 0.164 | 0.075 | 0.309
  Month 48 to end of study (N=8, 6, 3) | 0.000 | 0.000 | 0.000

4. Secondary Outcome: Percentage of Patients Relapse-free at the End of the Study
Description: Patients who did not experience any relapses confirmed by a neurologist during the study were regarded as relapse-free patients.
Time Frame: Baseline to the end of the study (up to 4 years)
Population: Core full analysis set (FAS): All patients who were randomized in the core study and received at least 1 dose of core study drug. The study became open-label with all patients receiving FTY720 0.5 mg/day (by 22-Feb- 2010).(approximately 22 months before study completion)
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Fingolimod 0.5 mg | Fingolimod 1.25 mg | Placebo-fingolimod
Number analyzed (Participants) | 57 | 54 | 57
Percentage of patients | 45.2 [26.87 to 61.95] | 62.1 [46.63 to 74.26] | 48.3 [33.29 to 61.77]

5. Secondary Outcome: Percentage of Patients Free From 3-month and 6-month Confirmed Disability Progression at Their Last Expanded Disability Status Scale (EDSS) Assessment
Description: Disability progression was measured by the EDSS score. A trained neurologist grades the multiple sclerosis (MS) disability of the patient on a scale of 0-5 (no to severe disability) in 8 Functional Systems (FS): Pyramidal, cerebellar, brainstem, sensory, bowel and bladder, visual, cerebral (or mental), and other. The EDSS score ranges from 0-10 (normal to dead) with higher scores indicating greater disability. A 3-month confirmed disability progression was defined as a 3-month sustained increase from baseline in the EDSS score, that is, every EDSS score obtained (scheduled or unscheduled) within 3-months after the first progression met the following progression criteria: One point (1) increase from baseline in patients with baseline EDSS score from 0 to 5.0; or half a point (0.5) increase in patients with baseline EDSS score of 5.5 or above. A 6-month confirmed disability progression was defined exactly the same except that the sustained progression had to last 6 months.
Time Frame: Baseline to the end of the study (up to 4 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Fingolimod 0.5 mg | Fingolimod 1.25 mg | Placebo-fingolimod
Number analyzed (Participants) | 57 | 54 | 57
Percentage of patients
  Free from 3-month confirmed disability progression | 74.3 [55.04 to 86.31] | 82.4 [67.73 to 90.87] | 90.6 [78.63 to 95.99]
  Free from 6-month confirmed disability progression | 87.1 [73.40 to 94.03] | 90.7 [76.94 to 96.44] | 92.3 [80.51 to 97.06]

6. Secondary Outcome: Change From Core Study Baseline in the Expanded Disability Status Scale (EDSS) Score
Description: as for outcome 5
Time Frame: Baseline to Months 12, 24, 36, 48, and end of study (up to 4 years)
Population: Core full analysis set (FAS): All patients who were randomized in the core study and received at least 1 dose of core study drug. • The study became open-label with all patients receiving FTY720 0.5 mg/day (by 22-Feb- 2010). (approximately 22 months before study completion)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fingolimod 0.5 mg | Fingolimod 1.25 mg | Placebo-fingolimod
Number analyzed (Participants) | 57 | 54 | 57
Units on a scale
  Month 12 (N=45, 43, 40) | -0.02 (0.464) | -0.02 (0.831) | -0.23 (0.800)
  Month 24 (N=42, 40, 35) | -0.12 (0.723) | -0.06 (1.033) | -0.21 (0.789)
  Month 36 (N=25, 21, 23) | 0.16 (1.441) | -0.07 (0.912) | -0.37 (0.678)
  Month 48 (N=3, 4, 1) | 1.17 (0.764) | -0.63 (0.946) | 0.00 (0.000)
  End of study (N=37, 36, 32) | 0.00 (1.225) | -0.17 (0.902) | -0.31 (0.830)

ADVERSE EVENTS:
Description: Extension safety population: All patients who received at least 1 dose of study drug in the extension study.
Arm/Group | Fingolimod 1.25 mg | Fingolimod 0.5 mg | Placebo-fingolimod 1.25 mg | Placebo-fingolimod 0.5 mg
Serious Adverse Events (participants affected / at risk) | 5/46 | 8/47 | 5/23 | 1/27
Other Adverse Events (participants affected / at risk) | 43/46 | 42/47 | 21/23 | 25/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod 1.25 mg (N=46) | Fingolimod 0.5 mg (N=47) | Placebo-fingolimod 1.25 mg (N=23) | Placebo-fingolimod 0.5 mg (N=27)
Bradycardia (Cardiac disorders) | 0 | 0 | 2 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0
Tooth impacted (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Eyeball rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0
Leukoencephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 0 | 1 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 1 | 0 | 0
Neuromyelitis optica (Nervous system disorders) | 0 | 0 | 0 | 1
Radiculitis (Nervous system disorders) | 0 | 0 | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Abortion induced (Surgical and medical procedures) | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod 1.25 mg (N=46) | Fingolimod 0.5 mg (N=47) | Placebo-fingolimod 1.25 mg (N=23) | Placebo-fingolimod 0.5 mg (N=27)
Leukopenia (Blood and lymphatic system disorders) | 5 | 2 | 1 | 4
Lymphopenia (Blood and lymphatic system disorders) | 8 | 6 | 3 | 2
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 3 | 0
Cataract (Eye disorders) | 2 | 3 | 1 | 2
Dry eye (Eye disorders) | 0 | 3 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3 | 0 | 2
Constipation (Gastrointestinal disorders) | 2 | 5 | 0 | 1
Dental caries (Gastrointestinal disorders) | 4 | 3 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 6 | 3 | 2 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Gastritis (Gastrointestinal disorders) | 2 | 3 | 0 | 1
Gingivitis (Gastrointestinal disorders) | 3 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 3 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 3 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 6 | 4 | 1 | 4
Seasonal allergy (Immune system disorders) | 1 | 1 | 2 | 0
Cystitis (Infections and infestations) | 7 | 3 | 1 | 2
Folliculitis (Infections and infestations) | 2 | 0 | 0 | 2
Herpes zoster (Infections and infestations) | 1 | 1 | 2 | 1
Influenza (Infections and infestations) | 6 | 3 | 3 | 2
Nasopharyngitis (Infections and infestations) | 28 | 29 | 12 | 15
Onychomycosis (Infections and infestations) | 1 | 1 | 0 | 2
Oral herpes (Infections and infestations) | 0 | 0 | 2 | 0
Pharyngitis (Infections and infestations) | 4 | 5 | 2 | 1
Sinusitis (Infections and infestations) | 3 | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 1 | 3 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 2
Blood triglycerides increased (Investigations) | 0 | 1 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 2 | 1
Liver function test abnormal (Investigations) | 8 | 6 | 9 | 7
Lymphocyte count decreased (Investigations) | 2 | 3 | 2 | 3
White blood cell count decreased (Investigations) | 3 | 2 | 2 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 5 | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 6 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 4 | 0 | 0
Headache (Nervous system disorders) | 3 | 8 | 3 | 1
Insomnia (Psychiatric disorders) | 2 | 4 | 1 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 3 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 4 | 3 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 4 | 1 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2
Hypertension (Vascular disorders) | 1 | 3 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.